CLINICAL TRIAL: NCT00465309
Title: Protective Ventilation With Carbon Dioxide (CO2) -Removal Technique in Patients With Adult Respiratory Distress Syndrome (ARDS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Collaborators: Regione Piemonte (Other)
Responsible Party: Marco Ranieri, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR60ANMA06
Record Dates: First submitted 2007-04-24; First posted 2007-04-25 (Estimated); Last update posted 2009-01-12 (Estimated); Status verified 2009-01

CONDITIONS: Adult Respiratory Distress Syndrome
Keywords: Respiratory Insufficiency; CO2 removal; protective ventilation; ARDS
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Insufficiency

INTERVENTIONS:
Procedure: protective ventilation with CO2 removal technique — In ARDS patients, presenting a Pplat ≥ 26 cmH2O, Vt was lowered (reaching a Pplat < 26) with CO2-removal veno-venous pump-driven bypass support for 48 consecutive hours with a pH > 7,30 or at least 72 hours from the beginning of the extracorporeal treatment.

SUMMARY:
30% of ARDS patients ventilated according to NIH protocol presents morphological (CT) and functional (Stress Index>1) conditions of hyperinflation even with Plateau pressure (Pplat) < 30 cmH2O; values of Pplat lower than 26 cmH2O were associated with more a condition of more protective ventilation.

In patients at risk of hyperinflation, use of alternative techniques such as CO2-removal my allow the reduction of Tidal Volume (Vt) and Pplat.

DETAILED DESCRIPTION:
Aim of the study was to verify the efficacy of CO2-removal technique in reducing Vt and consequently Pplat to obtain a Stress Index value equal to 1.

ELIGIBILITY:
Inclusion Criteria:

* ARDS patients with Pplat >= 26 during NIH protective ventilation protocol

Exclusion Criteria:

* Age < 18 years
* Brain injury and patients with intracranial pressure > 20 mmHg
* Pregnancy
* Immunodepressed patients
* Patients already enrolled in other trials
* Renal replacement therapy
* BMI > 40
* Contraindication anticoagulation treatment
* Morphological abnormalities of femoral veins
* NYHA III-IV
* Burns BSA>30%
* Hepatic failure (grade C Child)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-04; Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
pulmonary inflammatory mediator reduction | within the first 72 hours after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: V. M. Ranieri, MD, Study Director — University of Turin, Italy; P. Terragni, MD, Principal Investigator — University of Turin, Italy
Locations (2):
- Italy (2):
  - University of Turin, Department of Anesthesia and Intensive Care Medicine,S. G. Battista Hospital, Turin, Turin
  - University of Turin, Department of Anesthesia and Intensive Care Medicine, Turin

REFERENCES:
- [Background] Terragni PP, Rosboch G, Tealdi A, Corno E, Menaldo E, Davini O, Gandini G, Herrmann P, Mascia L, Quintel M, Slutsky AS, Gattinoni L, Ranieri VM. Tidal hyperinflation during low tidal volume ventilation in acute respiratory distress syndrome. Am J Respir Crit Care Med. 2007 Jan 15;175(2):160-6. doi: 10.1164/rccm.200607-915OC. Epub 2006 Oct 12. PMID 17038660